CLINICAL TRIAL: NCT04546100
Title: Effects of a Maternal-Infant Exercise Program on Body Composition, Stress, Fatigue, and Attachment in Postpartum Women：A Randomized Control Trial
Brief Title: Maternal-Infant Exercise Program on Body Composition, Stress, Fatigue, and Attachment in Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-2020-07-16
Record Dates: First submitted 2020-08-03; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Postpartum; Body Composition; Stress; Fatigue; Attachment
Keywords: postpartum; maternal-infant exercise program; body composition; stress; fatigue; attachment
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal-Infant Exercise Program (Experimental): In the postpartum period, give the intervention group "Maternal-Infant Exercise Program" and encourage them to do exercise. The "Parent-Child Exercise Program" can be divided into three stages. Videos will be provided in each stage. As time progresses during the three months, the parent-child exercise videos provided will have stronger intensity. The content includes general post-natal exercises (e.g., baby Lying on the mother's bed, raising legs or back of hands exercises, breast exercises; neck exercises; pelvic swinging exercises), aerobic exercises (e.g. walking with strollers, walking with baby on back), core exercises (e.g. kneeling balance, kneeling Push ups, stick exercises, modified side stick exercises) and hip and leg exercises (such as donkey kicks, side lifts), etc., with relaxing music during exercise.
  Interventions: Other: Maternal-Infant Exercise Program
- Regular postpartum exercise guidance (Placebo Comparator): Another group will receive "Regular postpartum exercise guidance". The guidance includes chest exercises, neck exercises, leg exercises, hip exercises, abdominal exercises, vagina contraction exercises, and uterine contraction exercises, starting from the third day after delivery to one month after delivery. The detail information will refer to the General Hospital of Tri-Services Provided the postpartum health education manual-postpartum exercise (p.8-10)
  Interventions: Other: Maternal-Infant Exercise Program

INTERVENTIONS:
Other: Maternal-Infant Exercise Program — "Maternal-Infant Exercise Program" can be divided into three videos stages. As time progresses during the three months, the parent-child exercise videos provided will have stronger intensity. The content includes general post-natal exercises (e.g., baby Lying on the mother's bed, raising legs or back of hands exercises, breast exercises; neck exercises; pelvic swinging exercises), aerobic exercises (e.g. walking with strollers, walking with baby on back), core exercises (e.g. kneeling balance, kneeling Push ups, stick exercises, modified side stick exercises) and hip and leg exercises (such as donkey kicks, side lifts), etc., with relaxing music during exercise.

SUMMARY:
The aim of this study is to explore the effectiveness of the intervention measures of the "Maternal-Infant Exercise Program" to improve the postpartum women's body composition, stress, fatigue and parent-child attachment.

DETAILED DESCRIPTION:
Background:

In Taiwan, more than 50% of maternal women will encounter obesity problems, because they have to take care of newborns, lack of proper exercise, and the traditional concept of confinement leads to excessive dietary supplementation, basal metabolic rate decline, and insufficient exercise. In addition to the physical changes after birth, women also face the change of the role of mothers. Caring for newborns is almost 24 hours on standby, gradually forming stress and fatigue. Stress may make postpartum women unable to perform the tasks of mothers. Makes postpartum women feel physiologically and psychologically uncomfortable. Both stress and fatigue have an adverse effect on their health, and are not conducive to parent-child attachment. However, early postpartum mothers and infants are almost inseparable. This period of attachment often affects infants' interpersonal relationships and emotions, if the relationship is not harmonious, may cause deviations in the baby's future behavior. Many studies have pointed out that moderate exercise can not only reduce the fatigue of postpartum women but also help to restore physical strength, help the recovery of organs and body, maintain physical health and weight management. However, busy with baby care and lack of continuous exercise often lead to postpartum women unable to reduce body weight. Therefore, this study hopes to develop a "Maternal-Infant Exercise Program" to improve the postpartum women's body composition, stress and fatigue, and to improve the attachment relationship between parents and their infants.

Purposes:

Explore the effectiveness of the intervention measures of the "Maternal-Infant Exercise Program" to improve the postpartum women's body composition, stress, fatigue and parent-child attachment.

Method:

In this study, a longitudinal and long-term follow-up randomized controlled trial study was adopted. The case was collected in a postpartum ward and an obstetrics and gynecology clinic of a medical center in the north Taiwan. The mothers who met the conditions for sample selection were selected as the research object. There are two different intervention modes (intervention group and control group), the intervention group is a Maternal-Infant Exercise Program, and the control group receives routine postpartum exercise nursing guidance. There are 50 people in each group. It is estimated that 100 healthy women with vagina postpartum will be collected. The questionnaires and physiological measurements are used to collect and aggregate the data. The main research variables are the Maternal-Infant Exercise Program, and the dependent variables are the postpartum women's body composition, stress, fatigue and parent-child attachment. The body composition of postpartum women is measured using a body fat meter, postpartum stress is measured using a Perceived Stress Scale(PSS), postpartum fatigue is measured using a Modified Fatigue Symptoms Checklist(MFSC), and the parent-child attachment relationship is measured using the Maternal Attachment Inventory(MAI). The two groups will collect data at one month, two months and three months after delivery, including body composition measurement and filling in each scale. The analysis method of the research data will use SPSS version 22.0 software, using chi-square test, independent sample t test , Pearson correlation, generalized estimation equations for discussion of results.

Result:

This study expects to understand the current status of postpartum women's body composition, stress, fatigue, and parent-child attachment. It is expected that parent-child exercise programs will improve postpartum women's body composition, as well as improve stress, fatigue, and enhance parent-child attachment.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum healthy women with vaginal delivery
2. No obstetric complications
3. Taiwanese, understand Chinese
4. Agreed to participate in the research after the explanation, and agreed to receive four questionnaire surveys
5. The baby's gestational weeks are more than 37 weeks and the birth weight is more than 2500 grams
6. The baby has no complications or no congenital abnormalities

Exclusion Criteria:

1. Four-degree laceration of the perineal wound
2. A history of serious medical and surgical diseases cannot perform exercise
3. Those who cannot cooperate with the implementation of the parent-child exercise program at least three days a week, 20-30 minutes each time
4. The infant must be hospitalized for observation after being evaluated by a doctor and cannot be discharged

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Composition- weight-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: weight(kg).
Body Composition- weight-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: weight(kg).
Body Composition- weight-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: weight(kg).
Body Composition- weight-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: weight(kg).
Body Composition- body mass index-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body mass index(kg/m2).
Body Composition- body mass index-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body mass index(kg/m2).
Body Composition- body mass index-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body mass index(kg/m2).
Body Composition- body mass index-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body mass index(kg/m2).
Body Composition- body fat-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body fat percentage(%).
Body Composition- body fat-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body fat percentage(%).
Body Composition- body fat-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data: body fat percentage(%).
Body Composition- body fat-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body fat percentage(%).
Body Composition- body water-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body water(%).
Body Composition- body water-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body water(%).
Body Composition- body water-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body water(%).
Body Composition- body water-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body water(%).
Body Composition- muscle mass-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:muscle mass(kg).
Body Composition- muscle mass-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:muscle mass(kg).
Body Composition- muscle mass-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:muscle mass(kg).
Body Composition- muscle mass-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:muscle mass(kg).
Body Composition- bone mass-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:bone mass(kg).
Body Composition- bone mass-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:bone mass(kg).
Body Composition- bone mass-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:bone mass(kg).
Body Composition- bone mass-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:bone mass(kg).
Body Composition- basal metabolic rate(BMR)-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:basal metabolic rate(kcal).
Body Composition- basal metabolic rate(BMR)-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:basal metabolic rate(kcal).
Body Composition- basal metabolic rate(BMR)-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:basal metabolic rate(kcal).
Body Composition- basal metabolic rate(BMR)-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:basal metabolic rate(kcal).
Body Composition- body age-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body age(age).
Body Composition- body age-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body age(age).
Body Composition- body age-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body age(age).
Body Composition- body age-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:body age(age).
Body Composition- Visceral fat-T1 | T1-baseline
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:visceral fat (level).
Body Composition- Visceral fat-T2 | T2-one month later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:visceral fat (level).
Body Composition- Visceral fat-T3 | T3-two months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:visceral fat (level).
Body Composition- Visceral fat-T4 | T4-three months later
  This study uses a body fat meter(TANITA BC-545N), and the Ministry of Health Medical Device Input No. 028886, which has been calibrated by the manufacturer before use. This device record data:visceral fat (level).

SECONDARY OUTCOMES:
Postpartum stress-T1 | T1-baseline
  The Perceived Stress Scale(PSS) has 14 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum stress.
Postpartum stress-T2 | T2-one month later
  The Perceived Stress Scale(PSS) has 14 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum stress.
Postpartum stress-T3 | T3-two months later
  The Perceived Stress Scale(PSS) has 14 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum stress.
Postpartum stress-T4 | T4-three months later
  The Perceived Stress Scale(PSS) has 14 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum stress.
Postpartum fatigue-T1 | T1-baseline
  The Modified Fatigue Symptoms Checklist(MFSC) has 10 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum fatigue.
Postpartum fatigue-T2 | T2-one month later
  The Modified Fatigue Symptoms Checklist(MFSC) has 10 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum fatigue.
Postpartum fatigue-T3 | T3-two months later
  The Modified Fatigue Symptoms Checklist(MFSC) has 10 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum fatigue.
Postpartum fatigue-T4 | T4-three months later
  The Modified Fatigue Symptoms Checklist(MFSC) has 10 questions on the scale. The questions use a response level of 0 to 4. The 0 point means never, 1 point means occasionally, 2 points means sometimes, 3 points means often,and 4 points means always. The higher the total score, the greater the postpartum fatigue.
Attachment-T1 | T1-baseline
  The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often. The higher the total score, the closer the maternal-infant attachment.
Attachment-T2 | T2-one month later
  The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often. The higher the total score, the closer the maternal-infant attachment.
Attachment-T3 | T3-two months later
  The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often. The higher the total score, the closer the maternal-infant attachment.
Attachment-T4 | T4-three months later
  The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often. The higher the total score, the closer the maternal-infant attachment.

CONTACTS AND LOCATIONS:
Locations (1):
- TSGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No